CLINICAL TRIAL: NCT02868476
Title: Long Period Observation of Biochemical Survey and Ultrasonography in Thyroid Diseases and Subclinical Thyroid Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201606056RINA
Record Dates: First submitted 2016-08-05; First posted 2016-08-16 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical and subclinical thyroid disease is usually used to describe patients with mild symptoms correlated to hyperthyroid or hypothyroid state. Therapeutic decision for clinical and subclinical thyroid dysfunction should be considered individually. But long term outcome for treatment of such functional and structural thyroid diseases had not been recorded delicately in Taiwan. Further investigations should be observed in the future.The purpose of this study is aiming for early prevention and detection the potential risk factors for thyroid diseases in Taiwan.

DETAILED DESCRIPTION:
Clinical and subclinical thyroid disease is usually used to describe patients with mild symptoms correlated to hyperthyroid or hypothyroid state. Thyroid ultrasonography could differentiate benign or malignant nodular lesion, together with fine needle aspiration cytology and surgical pathology. Thyrotropin (TSH, thyroid stimulating hormone) is the pivotal investigation in laboratory diagnosis to define subclinical thyroid diseases. An elevated TSH with normal free thyroxine and triiodothyronine levels in serum is defined to be subclinical hypothyroidism, and a subnormal TSH with normal thyroid hormone concentrations to be subclinical hyperthyroidism. Generally, the prevalence of subclinical hypothyroidism and hyperthyroidism were reported as 4% -10% & 1%-2% in general population, respectively. Although subclinical thyroid disease is prevalent, there is still no consensus for screening clinical and subclinical thyroid disease, including hyperthyroidism, hypothyroidism, nodular goiter and thyroid cancer. Under consideration of age, gender or familial history of autoimmune thyroid disease. However, screening for thyroid dysfunction should be considered in some high risk patients, including 1) elderly; 2) history of atrial fibrillation; 3) previous thyroid disease history; 4) other confirmed autoimmune diseases; 5) neck exposure of radiation (for example, nasopharyngeal cancer, post-radiation); 6) family history of probable autoimmune thyroid disease, and 7) pregnant state with prior thyroid disease history. Therapeutic decision for clinical and subclinical thyroid dysfunction should be considered individually. Therapeutic options will be anti-thyroid medications and/or radioactive iodine, and thyroidectomy could be considered with larger goiters for hyperthyroidism. For clinical and subclinical hypothyroidism, the therapeutic consideration should be aimed on reduction of progression to overt hypothyroidism, improving heart function, correction of dyslipidemia, and relieving senescence depressive mood. Thyroid ultrasonography will help us to keep long term observation of thyroid structural change. But long term outcome for treatment of such functional and structural thyroid diseases had not been recorded delicately in Taiwan. Further investigations should be observed in the future. We hope to check the relationship between various thyroid diseases and biochemical survey/ultrasonography. The purpose of this study is aiming for early prevention and detection the potential risk factors for thyroid diseases in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years old
* Thyroid diseases, including nodular goiter, hyperthyroidism, hypothyroidism and thyroid cancer (before or after operation), consecutive follow-up in outpatient department, and we expected to enroll 800 patients in one year, and follow-up with observation for 5 years.

Exclusion Criteria:

* N/A

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid diseases, age between 20 to 80 years old, consecutive follow-up in outptient department, and we expected to enroll 800 patients in one year, and follow-up with observation for 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Long Period Observation of Biochemical survey and Ultrasonography in Thyroid Diseases and Subclinical Thyroid Diseases | 5 years
  The study was designed as prospective pattern, and the investigators enrolled new patients with hyperthyroidism/hypothyroidism/nodular goiter/thyroid cancer with long period follow-up, then record thyroid change of thyroid function after treatment of anti-thyroid drugs or thyroid hormone replacement; the clinical outcome of nodular goiter with serial fine needle aspiration cytology and the correlation with thyroid ultrasonography, with the volume/echogenicity/vascularity of nodular goiters. Try to find the correlation of outcome (including how long will the anti-thyroid drugs be stopped without thyroid ablation, the natural course of benign nodular goiters without operation; or thyroid cancer recurrence, thyroid cancer, lymph nodes metastasis or distant metastasis, with surgery/radioactive iodine ablation/target therapy) with regular follow-up in outpatient department via time-dependent manner at least 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided